CLINICAL TRIAL: NCT06093243
Title: Women's Knowledge About Endometriosis
Acronym: Connaiss-Endo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_012_Connaiss-Endo
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Endometriosis
Keywords: Women; knowledge; endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "women of childbearing age" group: women of childbearing age with or without endometriosis
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection

SUMMARY:
In the world, 10% of women of childbearing age have endometriosis with diagnostic mostly between 25 and 30 years old.

Endometriosis is the leading cause of infertility in our country. A diagnosis delay of approximately 6.7 years is observed for endometriosis.

DETAILED DESCRIPTION:
The aim of the study will be to describe knowledge of women about endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* women older than 18
* women of childbearing age
* with or without gynecological history
* agreed to participate in the study

Exclusion Criteria:

None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women of childbearing age with or without endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
knowledge score on endometriosis symptoms | Day 0
  14 questions with yes/no answers, about symptoms of endometriosis (pain, nausea and vomiting, prolonged heavier period flow,…).
  A correct answer earns 1 point and a wrong answer earns 0 points. The knowledge score will therefore be between 0 and 14, the higher the score the better the knowledge.

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Reims Champagne Ardenne, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided